CLINICAL TRIAL: NCT01320189
Title: Dietary Protein Requirements and Caloric Over-consumption on Unbalanced Diets
Brief Title: Dietary Protein Requirements on Unbalanced Diets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Eveline Martens, PhD, Maastricht University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NL36167
Record Dates: First submitted 2011-03-16; First posted 2011-03-22 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Obesity; Overweight
Keywords: Energy intake; Protein requirement; Satiety; Protein leverage hypothesis
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Protein intake of 5 energy percent (Experimental)
  Interventions: Dietary Supplement: Differences in protein content of meals
- Protein intake of 15 energy percent (Experimental)
  Interventions: Dietary Supplement: Differences in protein content of meals
- Protein intake of 30 energy percent (Experimental)
  Interventions: Dietary Supplement: Differences in protein content of meals

INTERVENTIONS:
Dietary Supplement: Differences in protein content of meals — Differences in protein content (energy percent) of meals

SUMMARY:
The objective of this study is to determine ad libitum daily energy and protein intake, energy balance and appetite profile in response to protein/carbohydrate and fat ratio over 12 consecutive days, also as a function of age, gender, BMI and FTO polymorphisms.

DETAILED DESCRIPTION:
Following the protein leverage hypothesis, energy intake may be a derivative of protein intake. Therefore, in response to an unbalanced menu relative to the usual daily intake target, protein intake should be prioritized. Individuals may over-consume carbohydrate and fat of a menu containing a lower ratio of protein to carbohydrate and fat until the daily intake target amount of protein is ingested, and not the target of total energy intake because of a deficit of protein intake. In contrast, individuals may under-consume energy when the menu has an increased protein to carbohydrate and fat ratio. The protein leverage hypothesis requires evidence for why protein intake is more important than carbohydrate or fat in relation to food intake regulation.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-35 kg/m2
* age between 18-70 years
* healthy
* non-smoking
* not using a more than moderate amount of alcohol (> 10 consumptions/wk)
* weight stable (weight change < 3 kg during the last 6 months)
* not using medication or supplements except for oral contraceptives in women

Exclusion Criteria:

* not healthy
* smoking
* using a more than moderate amount of alcohol
* not being weight stable
* using medication or supplements except for oral contraceptives in women
* do not meet the criteria for BMI and age
* pregnant or lactating
* allergic for the used food items

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2011-05; Primary Completion 2012-02 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
energy intake | 12 consecutive days
protein intake | 12 consecutive days
energy balance | 12 consecutive days
appetite profile | 12 consecutive days

CONTACTS AND LOCATIONS:
Overall Officials: Margriet S. Westerterp-Plantenga, Prof. dr., Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Department of Human Biology, Nutrition and Toxicology Research Institute Maastricht (NUTRIM), Maastricht, Maastricht, Netherlands

REFERENCES:
- [Result] Simpson SJ, Raubenheimer D. Obesity: the protein leverage hypothesis. Obes Rev. 2005 May;6(2):133-42. doi: 10.1111/j.1467-789X.2005.00178.x. PMID 15836464
- [Result] Sorensen A, Mayntz D, Raubenheimer D, Simpson SJ. Protein-leverage in mice: the geometry of macronutrient balancing and consequences for fat deposition. Obesity (Silver Spring). 2008 Mar;16(3):566-71. doi: 10.1038/oby.2007.58. Epub 2008 Jan 17. PMID 18239565
- [Result] Weigle DS, Breen PA, Matthys CC, Callahan HS, Meeuws KE, Burden VR, Purnell JQ. A high-protein diet induces sustained reductions in appetite, ad libitum caloric intake, and body weight despite compensatory changes in diurnal plasma leptin and ghrelin concentrations. Am J Clin Nutr. 2005 Jul;82(1):41-8. doi: 10.1093/ajcn.82.1.41. PMID 16002798
- [Result] Leidy HJ, Tang M, Armstrong CL, Martin CB, Campbell WW. The effects of consuming frequent, higher protein meals on appetite and satiety during weight loss in overweight/obese men. Obesity (Silver Spring). 2011 Apr;19(4):818-24. doi: 10.1038/oby.2010.203. Epub 2010 Sep 16. PMID 20847729
- [Derived] Martens EA, Tan SY, Mattes RD, Westerterp-Plantenga MS. No protein intake compensation for insufficient indispensable amino acid intake with a low-protein diet for 12 days. Nutr Metab (Lond). 2014 Aug 20;11:38. doi: 10.1186/1743-7075-11-38. eCollection 2014. PMID 25183991
- [Derived] Martens EA, Lemmens SG, Westerterp-Plantenga MS. Protein leverage affects energy intake of high-protein diets in humans. Am J Clin Nutr. 2013 Jan;97(1):86-93. doi: 10.3945/ajcn.112.046540. Epub 2012 Dec 5. PMID 23221572